CLINICAL TRIAL: NCT04197193
Title: Monitoring Antioxidant/Redox Status and Replenishing Nitrogen & Sulfur-based Nutrients to Enhance Resilience at Concordia (MARS-C): Understanding Integrated Stress Signalling
Brief Title: Monitoring Antioxidant/Redox Status at Concordia (MARS-C)
Acronym: MARS-C
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Southampton (Other)
Collaborators: European Space Agency (Other)
Responsible Party: Sponsor
Other Study IDs: 49348
Record Dates: First submitted 2019-12-04; First posted 2019-12-13 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2024-01

CONDITIONS: Oxidative Stress

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The European Space Agency (ESA) runs a research centre in Antarctica as an earth-based model for long duration deep-space missions. Just like astronauts travelling into space, crew-members overwintering at this Concordia base are exposed to a number of extreme environmental stressors; including high altitude (approximately 3800m); extreme cold; long periods of 24 hour darkness or daylight; and complete isolation. The investigators will recruit up to 30 over-wintering crew members working at this station for ESA over a 2 year period and observe how their bodies adapt and respond to the stress of living and working in this environment. The investigators will collect blood, saliva and urine samples, together with ultrasound images of muscle mass and grip strength measurements at regular intervals throughout their deployment to Antarctica. These samples will be transported back to Southampton to be analysed for biochemical levels of stress. During the final month of their stay, all participants will be randomised to receive a daily nutritional drink which is either high or low in targeted dietary supplements. Following similar studies that the investigators has successfully performed over shorter durations at high altitudes previously, they hypothesise that levels of stress experienced in extreme environments such as Antarctica or deep space can be reduced with targeted nutritional supplementation. These findings may become important to members of the general public as commercial aviation moves increasingly towards using low space-orbital vehicles to drastically reduce international travel times over the coming decade.

ELIGIBILITY:
Inclusion Criteria:

* Adult
* Member of Concordia station over-wintering crew
* Able to give written informed consent
* Fluent in either English, French or Italian

Exclusion Criteria:

* Participating in another interventional research study during the deployment to Concordia

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Over-wintering members of Concordia crew
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2022-10-03 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Hand grip strength | up to 10 months
  Forearm muscle / grip strength recorded non-invasively using a hand grip dynamometer

SECONDARY OUTCOMES:
Muscle mass | up to 10 months
  cross sectional forearm muscle area recorded a standardised way using medical ultrasound
Oxidative stress | up to 10 months
  Nitrate, nitrite, nitroso species, FRAP, TFTs, glutathione ratios, 8-isoprostane,
Lake Louise Score 2018 | up to 10 months
  A validated measure of altitude related symptoms and illness which scores symptoms across 4 different domains: headache, GI disturbance, fatigue & dizziness. Each is scored from 0 - 3 (for no symptoms to very debilitating respectively) and a total score of 3 or more including at headache symptoms is required for a positive diagnosis of Acute Mountain Sickness

CONTACTS AND LOCATIONS:
Overall Officials: Martin Feelisch, PhD, Principal Investigator — University of Southampton
Locations (1):
- University of Southampton, Southampton, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided